CLINICAL TRIAL: NCT06794333
Title: Comparative Efficacy of Trans-Perineal Laser Ablation Vs Water Vapor Ablation for Benign Prostatic Hyperplasia: a Single Center Randomized Controlled Trial
Brief Title: Single Center Comparative Trial of Trans-Perineal Laser Ablation Vs Water Vapor Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, ALESSANDRO ZUCCHI, Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPIT_2; PROGETTO SMART REGIONE TOSCANA (Other: REGIONE TOSCANA)
Record Dates: First submitted 2024-10-16; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-05

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; MISTs; LUTS; Rezum Vapor Therapy; Transperineal Laser Ablation
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transperineal Laser Ablation (Experimental): Treatments are performed with the combined EchoLaser EVO system (Elesta SpA - Calenzano, FI). The EchoLaser EVO consists of the Echolaser X4, a multi-source laser system with a wavelength of 1064 nm, and the Echolaser Smart Interface (ESI).
  The procedure are performed with the patient in the lithotomy position. Local anesthesia of the perineal region and periprostatic block with lidocaine is administered under ultrasound guidance. A catheter is placed during the irradiation to allow continuous irrigation of the urethra with saline solution, protecting the urethra from temperature rise. The Echolaser Smart Interface, defines: the number and positioning of fibers, the optimal dose, and the need for multiple pullbacks. 2 to 4 21G needles are inserted simultaneously (1 or 2 per lobe) in the peri-urethral area via transperineal ultrasound guidance. A 300-micron optical fiber will be placed in each needle. Each treatment delivers a maximum energy of 1800 J per fiber with a power of 3-5 W.
  Interventions: Procedure: Transperineal laser Ablation
- Rezum Vapor Therapy (Active Comparator): The treatment involves the insertion of a radiofrequency needle into the prostate tissue and the emission of water vapor.
  Treatment under local anesthesia/sedation. Treatment planning using the REZUM device, with the number of injections proportional to the recommended therapeutic scheme based on prostate volume (1 injection every centimeter starting 1 cm below the bladder neck and 1 cm in front of the verumontanum).
  Water vapor emission for 9-second intervals with a maximum of 9 applications per patient.
  Three-way bladder catheter to decrease local temperature. The bladder catheter will be removed 15 days after patient discharge. Regarding the REZUM, it is a system that uses sterile single-use handpieces available within the company, where a special optics is inserted for direct visualization. The handpiece features a device that allows the manual insertion of a needle into the prostate, from which water vapor is emitted for the described treatment.
  Interventions: Procedure: Rezum Vapor Therapy

INTERVENTIONS:
Procedure: Transperineal laser Ablation — Treatments are performed with the combined EchoLaser EVO system (Elesta SpA - Calenzano, FI). The EchoLaser EVO consists of the Echolaser X4, a multi-source laser system with a wavelength of 1064 nm, and the Echolaser Smart Interface (ESI). The procedure are performed with the patient in the lithotomy position. Local anesthesia of the perineal region and periprostatic block with lidocaine is administered under ultrasound guidance. A catheter is placed during the irradiation to allow continuous irrigation of the urethra with saline solution, protecting the urethra from temperature rise. The Echolaser Smart Interface, defines: the number and positioning of fibers, the optimal dose, and the need for multiple pullbacks. 2 to 4 21G needles are inserted simultaneously (1 or 2 per lobe) in the peri-urethral area via transperineal ultrasound guidance. A 300-micron optical fiber will be placed in each needle. Each treatment delivers a maximum energy of 1800 J per fiber with a power of 3-5 W.
  Other Names: EchoLaser EVO
  Arms: Transperineal Laser Ablation
Procedure: Rezum Vapor Therapy — The treatment involves the insertion of a radiofrequency needle into the prostate tissue and the emission of water vapor. Treatment under local anesthesia/sedation. Treatment planning using the REZUM device, with the number of injections proportional to the recommended therapeutic scheme based on prostate volume (1 injection every centimeter starting 1 cm below the bladder neck and 1 cm in front of the verumontanum). Water vapor emission for 9-second intervals with a maximum of 9 applications per patient. Three-way bladder catheter to decrease local temperature. The bladder catheter will be removed 15 days after patient discharge. Regarding the REZUM, it is a system that uses sterile single-use handpieces available within the company, where a special optics is inserted for direct visualization. The handpiece features a device that allows the manual insertion of a needle into the prostate, from which water vapor is emitted for the described treatment.
  Arms: Rezum Vapor Therapy

SUMMARY:
The primary aim of this clinical trial is to determine whether one of the two methods under investigation, TPLA or WVA, is superior in the treatment of BPH. Additionally, as a secondary objective, the study seeks to evaluate the potential superiority of one method over the other concerning the sexual parameters of treated participants, assessed using the International Index of Erectile Function 5 (IIEF5) and the Male Sexual Health Questionnaire - Ejaculatory Dysfunction (MSHQ-EJ).

The researchers will compare the two methods under investigation (TPLA and WVA) to assess the potential superiority of one over the other.

Participants will:

* be randomized 1:1 between the two techniques and will undergo treatment at time 0;
* undergo follow-up including uroflowmetry and assessment of the International Prostate Symptoms Score (IPSS), IIEF5, and MSHQ-EJ questionnaires at 3, 6, and 12 months.

DETAILED DESCRIPTION:
Therapeutic options for the treatment of benign prostatic hyperplasia (BPH) encompass a wide range of both pharmacological and surgical approaches. BPH is an age-related condition that increasingly affects relatively younger individuals, starting from the age of 50.

Pharmacological therapy primarily involves medications that can alleviate symptoms but do not cure or lead to a regression of the prostate gland enlargement over time.

Surgical therapy aims to reduce the degree of obstruction, and in most cases, it can result in significant alterations in sexual function, such as inducing retrograde ejaculation or causing erectile dysfunction. These side effects are more common with the use of classical treatment methods, whose clinical value is widely recognized and confirmed by clinical evidence reported in international guidelines (EAU Guidelines, 2021 edition).

The classical surgical treatment methods include the removal of the adenoma (benign hyperplastic part of the prostate gland) through open surgery, transurethral resection (TURP), laser ablation with en bloc removal (holmium and thulium lasers), or direct cavitation (green light laser). These classical methods typically require hospital admission with a stay of three days or more, depending on the extent of postoperative bleeding and the risk of post-surgical obstructive complications (bladder clots).

On the other hand, some minimally invasive and innovative methods can reduce the symptoms caused by the disease while preserving the patient's sexual function. These techniques also allow for treatment without hospitalization or, at most, in a outpatients setting, utilizing local anesthesia or sedation and presenting a low risk of bleeding or other complications. Specifically, the minimally invasive technologies aim for thermal ablation of the hyperplastic tissue without cavitation. This approach results in longer healing times and clinical improvement, as they are dependent on cellular apoptosis, tissue necrosis, and spontaneous gland remodeling, which occur in the months following treatment, thus not producing immediate visible or effective results.

These methods include Rezum (WVA), I-Tind, and SoracteLite trans-perineal laser ablation (TPLA). All of these minimally invasive methods have been extensively validated by clinical studies and scientific evidence.

SoracteLite-TPLA increases the temperature of the treated tissue through the absorption of laser radiation delivered to the targeted tissue by very thin optical fibers inserted perineally. Exposure to high temperatures causes coagulative necrosis of the tissues. In contrast, WVA involves the transurethral injection of water vapor through a radiofrequency needle. The local temperature increase generated by radiofrequency and water vapor leads to progressive tissue necrosis, reducing the size of the prostate adenoma and significantly improving urinary flow.

It is also logical that the use of minimally invasive methods allows for treating a larger number of patients with a lower risk of complications, although with an apparently reduced effectiveness in deobstruction compared to classical methods. The economic and social advantages are further highlighted by the faster resolution of waiting lists and greater psychological acceptance by the patient, due to the preservation of certain sexual functions and the reduced personal burden associated with the complex system of hospitalization/anesthesia/surgery/outcomes.

The primary objective is to evaluate the efficacy of TPLA vs WVA treatment at 3, 6, and 12 months in patients with BPH in terms of improvement in uroflowmetry parameters and symptoms. Specifically, the uroflowmetry parameters analyzed include maximum flow (Qmax), average flow (Qmed), and post-void residual (PVR). For symptom assessment, the IPSS questionnaire will be used.

The secondary objective includes evaluating the impact of these methods on the sexual health of treated participants through the IIEF5 and MSHQ-EJ questionnaires, which will be administered at 3, 6, and 12 months.

All participants will therefore undergo follow-up at 3, 6, and 12 months, during which they will undergo uroflowmetry with recording of Qmax, Qmed, and PVR parameters, as well as administration of the IPSS, IIEF5, and MSHQ-EJ questionnaires. This is a single-center randomized clinical trial in which participants are randomized 1:1 into the two treatment arms by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* PSA levels under 4 ng/ml (if PSA is over 4 ng/ml, a multiparametric prostate magnetic resonance will be performed; if a lesion with a PIRADS score over 2 is detected, a prostate biopsy will be conducted);
* Post void residual (PVR) over 50 ml;
* Maximum flow (Qmax) under 15 ml/s;
* IPSS score over 7;
* The possibility of undergoing transrectal ultrasound to assess the size of the prostate and prostate adenoma;
* Negative urinary culture.

Exclusion Criteria:

* Diabetes;
* Overactive or Underachieve bladder;
* Contraindications for performing MRI or prostate biopsy in cases where PSA is over 4 ng/ml;
* Intolerance to transrectal ultrasound;
* Intolerance or allergy to local anesthetics.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Improvement of Urodynamics parameters after 3 and 12 Months of Follow up | up to 12 months
  After 3,6 and 12 months of follow-up, uroflowmetry will be conducted to assess improvements in urinary maximum flow (Qmax: ml/sec) and average flow (Qmed: ml/sec). Milliliters and seconds will be combined to calculate and report Qmax and Qmed.
Improvement in post voided residual | up to 12 months
  After 3,6 and 12 months of follow-up, uroflowmetry will be conducted to assess improvements post voided residual (PVR: ml). Milliliters will be used to report PVR.
Improvement in International Prostate Symptoms Score | up to 12 months
  After 3,6 and 12 months of follow-up International Prostate Symptom Score (IPSS) questionnaire will be administered to all participants to evaluate changes in subjective symptoms and quality of life (Lower IPSS values indicate an improvement in the symptoms reported by the patient). The IPSS ranges from 0 to 35, with scores interpreted as follows: 0-7 indicates mild symptoms, 8-19 indicates moderate symptoms, and 20-35 indicates severe symptoms.

SECONDARY OUTCOMES:
Postoperative complications | up to 3 months
  Evaluate the incidence of postoperative complications according to Calvin Dindo Classification.
  The Clavien-Dindo classification categorizes complications related to a surgical procedure on a scale from 1 to 5. The severity of the complication increases with higher Clavien-Dindo scores.
Prostate Specific Antigen (PSA) value | up to 12 months
  To evaluate the PSA levels at 3,6 and 12 months. PSA will be reported by combining nanograms and milliliters (ng/ml).
sexual outcomes | up to 12 months
  To assess the impact of the procedures on penile erection, we will use the International Index of Erectile Function (IIEF5) questionnaire.
  The two questionnaires do not have units of measurement; they are expressed in absolute numbers. Higher IIEF5 values indicate better erectile function.
  The IIEF-5 score ranges from 0 to 25. Scores of 22 to 25 indicate normal erectile function, while scores of 17 to 21 suggest mild erectile dysfunction. Scores between 12 and 16 indicate mild-to-moderate dysfunction, 8 to 11 moderate dysfunction, and scores below 7 indicate severe erectile dysfunction.
sexual outcomes | up to 12 months
  To assess the impact of the procedures on anterograde ejaculatory function, we will use the Male Sexual Health Questionnaire - Ejaculation Disfunction (MSHQ-EJD).
  Higher scores reflect better ejaculatory function, with the questionnaire ranging from 0 to 15. Additionally, a final question, scored from 0 to 5, assesses the difficulty experienced by the patient during ejaculation. For this specific question, higher scores correspond to greater levels of difficulty reported (0: no difficulty, 5: extremely bothered).

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Zucchi, Professor, Study Chair — University of Pisa
Locations (1):
- University of Pisa, Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Riel LAMJG, van Kollenburg RAA, Vis AN, van Leeuwen PJ, de Reijke TM, de Bruin DM, Oddens JR. Safety and Feasibility of Soractelite Transperineal Focal Laser Ablation for Prostate Cancer and Short-term Quality of Life Analysis from a Multicenter Pilot Study. Eur Urol Open Sci. 2022 Apr 2;39:48-54. doi: 10.1016/j.euros.2022.02.012. eCollection 2022 May. PMID 35528781
- [Background] McVary KT, Roehrborn CG. Three-Year Outcomes of the Prospective, Randomized Controlled Rezum System Study: Convective Radiofrequency Thermal Therapy for Treatment of Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia. Urology. 2018 Jan;111:1-9. doi: 10.1016/j.urology.2017.10.023. Epub 2017 Nov 6. PMID 29122620
- [Background] Patelli G, Ranieri A, Paganelli A, Mauri G, Pacella CM. Transperineal Laser Ablation for Percutaneous Treatment of Benign Prostatic Hyperplasia: A Feasibility Study. Cardiovasc Intervent Radiol. 2017 Sep;40(9):1440-1446. doi: 10.1007/s00270-017-1662-9. Epub 2017 May 4. PMID 28474112
- [Background] Pacella CM, Patelli G, Iapicca G, Manenti G, Perretta T, Ryan CP, Esposito R, Mauri G. Transperineal laser ablation for percutaneous treatment of benign prostatic hyperplasia: a feasibility study. Results at 6 and 12 months from a retrospective multi-centric study. Prostate Cancer Prostatic Dis. 2020 Jun;23(2):356-363. doi: 10.1038/s41391-019-0196-4. Epub 2019 Dec 11. PMID 31827239
- See also: Related Info — https://www.elesta-echolaser.com